CLINICAL TRIAL: NCT02592252
Title: Cluster Randomised Controlled Trial to Assess the Impact of Combined Microfinance and Gender Training for Women and Gender Training for Women and Their Male Partners in Reducing Intimate Partner Violence
Brief Title: Impact of Microfinance and Participatory Gender Training for Women in Reducing Intimate Partner Violence
Acronym: MAISHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Mwanza Intervention Trials Unit (Other); National Institute for Medical Research, Tanzania (Other Government); Bangladesh Rural Advancement Committee (Other); EngenderHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QA430
Record Dates: First submitted 2015-08-13; First posted 2015-10-30 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Maltreatment by Spouse or Partner

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Microfinance + gender training (Experimental): Microfinance + 10 sessions of participatory gender training
  Interventions: Behavioral: Participatory gender training; Other: Microfinance
- Microfinance only (Experimental): Receive microfinance only
  Interventions: Other: Microfinance
- Gender training only (Experimental): 10 sessions of participatory gender training for women and their male partners
  Interventions: Behavioral: Participatory gender training
- No intervention (No Intervention): No microfinance or participatory gender training

INTERVENTIONS:
Behavioral: Participatory gender training — 10 sessions of participatory gender training
  Arms: Gender training only; Microfinance + gender training
Other: Microfinance — Microfinance loan
  Arms: Microfinance + gender training; Microfinance only

SUMMARY:
Violence against women and girls is increasingly recognized as a major global public health and development concern. However, evidence on what forms of intervention should be prioritised is severely lacking. A cluster randomized controlled trial (The Intervention with Microfinance for AIDS & Gender Equity - IMAGE Project) in rural South Africa combined a group-based microfinance intervention with a participatory gender and HIV training curriculum for loan participants and showed that, over a two-year period, levels of physical and/or sexual partner violence experienced by participants in the past year were reduced by 55%.

The overall goal of the current study is to design and implement a cluster randomized controlled trial to assess the impact on intimate partner violence of: 1) combining participatory gender training with microfinance for women in existing microfinance loan groups, and 2) a participatory gender training programme for women (not receiving microfinance) and their male partners.

ELIGIBILITY:
Inclusion Criteria:

Arms 1 and 2 - microfinance loan groups:

1. there are between 15 and 30 active members in the group
2. less than 25% of the women have been members for less than one year
3. there is a good attendance (repayment) record
4. a minimum of 70% of active members consent to take part in the study

Arms 3 and 4, women who:

1. are aged 20-50 years
2. are not formally employed, i.e. either self-employed or not currently working
3. have been resident in Mwanza for at least two years
4. have not been a member of a microfinance loan group in the past 12 months
5. are fluent in Swahili
6. have consented to take part in the study.

Exclusion Criteria:

None

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2640 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Past 12 months exposure to intimate partner violence | 24 months post-intervention
  Exposure to intimate partner violence will be assessed using the WHO Multi-country Study on Women's Health and Domestic Violence against Women questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Mawanza Intervention Trials Unit, Mwanza, Tanzania

REFERENCES:
- [Derived] Abramsky T, Guadarrama DS, Kapiga S, Mtolela G, Madaha F, Lees S, Harvey S. Pathways to reduced physical intimate partner violence among women in north-western Tanzania: Evidence from two cluster randomised trials of the MAISHA intervention. PLOS Glob Public Health. 2023 Nov 13;3(11):e0002497. doi: 10.1371/journal.pgph.0002497. eCollection 2023. PMID 37956111
- [Derived] Abramsky T, Harvey S, Mosha N, Mtolela G, Gibbs A, Mshana G, Lees S, Kapiga S, Stockl H. Longitudinal inconsistencies in women's self-reports of lifetime experience of physical and sexual IPV: evidence from the MAISHA trial and follow-on study in North-western Tanzania. BMC Womens Health. 2022 Apr 15;22(1):120. doi: 10.1186/s12905-022-01697-y. PMID 35428296
- [Derived] Harvey S, Abramsky T, Mshana G, Hansen CH, Mtolela GJ, Madaha F, Hashim R, Kapinga I, Watts C, Lees S, Kapiga S. A cluster randomised controlled trial to evaluate the impact of a gender transformative intervention on intimate partner violence against women in newly formed neighbourhood groups in Tanzania. BMJ Glob Health. 2021 Jul;6(7):e004555. doi: 10.1136/bmjgh-2020-004555. PMID 34301673
- [Derived] Kapiga S, Harvey S, Mshana G, Hansen CH, Mtolela GJ, Madaha F, Hashim R, Kapinga I, Mosha N, Abramsky T, Lees S, Watts C. A social empowerment intervention to prevent intimate partner violence against women in a microfinance scheme in Tanzania: findings from the MAISHA cluster randomised controlled trial. Lancet Glob Health. 2019 Oct;7(10):e1423-e1434. doi: 10.1016/S2214-109X(19)30316-X. PMID 31537372
- [Derived] Abramsky T, Lees S, Stockl H, Harvey S, Kapinga I, Ranganathan M, Mshana G, Kapiga S. Women's income and risk of intimate partner violence: secondary findings from the MAISHA cluster randomised trial in North-Western Tanzania. BMC Public Health. 2019 Aug 14;19(1):1108. doi: 10.1186/s12889-019-7454-1. PMID 31412825
- [Derived] Harvey S, Lees S, Mshana G, Pilger D, Hansen C, Kapiga S, Watts C. A cluster randomized controlled trial to assess the impact on intimate partner violence of a 10-session participatory gender training curriculum delivered to women taking part in a group-based microfinance loan scheme in Tanzania (MAISHA CRT01): study protocol. BMC Womens Health. 2018 Apr 2;18(1):55. doi: 10.1186/s12905-018-0546-8. PMID 29609568
- [Derived] Kapiga S, Harvey S, Muhammad AK, Stockl H, Mshana G, Hashim R, Hansen C, Lees S, Watts C. Prevalence of intimate partner violence and abuse and associated factors among women enrolled into a cluster randomised trial in northwestern Tanzania. BMC Public Health. 2017 Feb 14;17(1):190. doi: 10.1186/s12889-017-4119-9. PMID 28193198